CLINICAL TRIAL: NCT02858674
Title: Health Information Technology in Heart Failure Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14-01555
Record Dates: First submitted 2016-08-03; First posted 2016-08-08 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Alerting Mechanism (Experimental): Traditional Pop Up Alert used in Epic
  Interventions: Other: Pop Up Interruption Alert
- Passive Alerting Mechanism (Active Comparator): Noninterruptive alert that sits in the checklist
  Interventions: Other: Side Bar Non Interruptive Provider Checklist

INTERVENTIONS:
Other: Pop Up Interruption Alert — Traditional Pop Up Alert used in Epic
  Arms: Active Alerting Mechanism
Other: Side Bar Non Interruptive Provider Checklist — Noninterruptive alert that sits in the checklist
  Arms: Passive Alerting Mechanism

SUMMARY:
The objective of this proposal is to develop, implement, and test the effectiveness of a computerized clinical decision support system for hospitalized patients with heart failure.

Aim 1: Develop an electronic health record (EHR) based search method that uses both structured data and natural language processing of unstructured text to identify hospitalized patients with heart failure while they are still in the hospital.

Aim 2: Develop and test the usability of an electronic health record (EHR) based clinical decision support system (CDSS) to support delivery of evidence-based care to hospitalized heart failure patients using human computer interaction methods.

Aim 3: Assess the effect of an electronic health record (EHR) based clinical decision support system (CDSS) on processes of care for heart failure patients who are hospitalized for other causes. As part of the evaluation, we will test two implementation strategies, one of which will introduce the CDSS as an interruptive alert to providers, the second of which will introduce the CDSS as part of a provider checklist that exists on the side of the screen for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized 2 years prior and 18 months after the time of implementation of the Computerized clinical decision support systems (CDSS) in the (Electronic Health Record (EHR).

Exclusion Criteria:

* Patients on the obstetrical service, who died during hospitalization, or on hospice care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 958 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Percent of Patients with a Secondary Diagnoses of Heart Failure | 90 Days
  These patients will also have had of left ventricular function (LV) Assessment either prior to or during the hospitalization or planned for post discharge
Percentage of patients with a secondary diagnosis of heart failure and LV systolic dysfunction who have been prescribed an Angiotensin-converting enzyme (ACE) inhibitor or Angiotensin II receptor blockers (ARB) | 90 Days

CONTACTS AND LOCATIONS:
Overall Officials: Saul Blecker, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Blecker S, Austrian JS, Horwitz LI, Kuperman G, Shelley D, Ferrauiola M, Katz SD. Interrupting providers with clinical decision support to improve care for heart failure. Int J Med Inform. 2019 Nov;131:103956. doi: 10.1016/j.ijmedinf.2019.103956. Epub 2019 Sep 4. PMID 31525580